CLINICAL TRIAL: NCT00750893
Title: Safety of GlaxoSmithKline Biologicals' Oral Live Attenuated Human Rotavirus Vaccine, Rotarix or Rotarix Liquid Formulation (Oral Suspension or Prefilled Syringe) When Administered According to the Prescribing Information in Korea
Brief Title: Evaluation of Reactogenicity and Safety of GSK Biologicals' Rotarix (Human Rotavirus Vaccine) in Infants
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111700
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Infections, Rotavirus
Keywords: Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — RIX4414 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rotarix Group: Subjects who received 2 oral doses of Rotarix. The first dose was administered before the age of 6 weeks and the second one at least 4 weeks after, preferably before the age of 16 weeks. The 2 doses had to be given before 24 weeks of age.
  Interventions: Biological: Rotarix or Rotarix liquid formulation

INTERVENTIONS:
Biological: Rotarix or Rotarix liquid formulation — GSK Biologicals' oral live attenuated human rotavirus (HRV) vaccine (oral suspension or prefilled syringe).

SUMMARY:
This protocol posting deals with objectives and outcome measures of the primary phase at one month post-Dose 2. This Post Marketing Surveillance (PMS) will collect safety data on the use of human rotavirus vaccine in at least 3000 evaluable infants in Korea. This study involves male or female infants from the age of 6 weeks at the time of the first vaccination. The vaccination course must be completed by the age of 24 weeks.

DETAILED DESCRIPTION:
The protocol posting has been amended to reflect the two new vaccine presentations that have been launched in Korea. The current PMS will thus collect safety information from subjects who have received either Rotarix or Rotarix liquid formulation (oral suspension or prefilled syringe) in the course of their routine clinical practice according to the prescribing information in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Infants who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the PMS.
* A male or female infant from the age of 6 weeks at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the infant.

Exclusion Criteria:

• At the time of PMS entry, the contraindications and precautions of use indicated in the prescribing information should be checked and the infant must not be included in the PMS if there is any contraindication. Any changes in the locally approved Prescribing Information must be implemented immediately.

Ages: 6 Weeks to 24 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants aged at least 6 weeks will be administered two doses of Rotarix or Rotarix liquid formulation (oral suspension or prefilled syringe) orally as per the prescribing information in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 3111 (Actual)
Dates: Start 2008-09-02 (Actual); Primary Completion 2013-06-15 (Actual); Study Completion 2013-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shin SM, Kim CS, Karkada N, Liu A, Jayadeva G, Han HH. Post-marketing safety surveillance conducted in Korea (2008-2013) following the introduction of the rotavirus vaccine, RIX4414 (Rotarix). Hum Vaccin Immunother. 2016 Oct 2;12(10):2590-2594. doi: 10.1080/21645515.2016.1189046. Epub 2016 Aug 5. PMID 27494163
- See also: Full CSR posting. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=111700&attachmentIdentifier=979ab41f-0b4f-477f-b016-40716584106a&fileName=gsk-111700-clinical-study-report-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This post marketing study (PMS) covered a period of 6 consecutive years. Results were presented for Years 1, 2, 3, 4, 5 (Year [Y] 1 & Y2 data combined and presented at the Y2 time point and Y3 & Y4 data combined and presented at the Y4 time point) along with consolidated surveillance data from Y1- Y6 timepoint.
Pre-assignment Details: Consolidated participant flow and baseline measure data were given for Years 1 to 6 time point in order to account for all the subjects participating in this study.
Period: Overall Study
Arm/Group | Rotarix Group
Started | 3111
Completed | 2569
Not Completed | 542
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 510
Not completed — Other | 17

BASELINE CHARACTERISTICS:
Arm/Group | Rotarix Group
Number analyzed (Participants) | 3111
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 9.6 (2.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1525
  Male | 1586
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 3107
  Chinese | 2
  Japanese | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include cough, diarrhoea, irritability, loss of appetite, temperature and vomiting.
Time Frame: During the 8-day follow-up period after each vaccine dose for Year 1 & Year 2 study period
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one dose of Rotarix vaccine administration documented and for whom data were available at Year 1 and Year 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group
Number analyzed (Participants) | 876
Participants
  Cough | 204
  Diarrhoea | 50
  Irritability | 405
  Loss of appetite | 259
  Temperature | 135
  Vomiting | 200

2. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs) During the 31-day Follow-up Period After Each Vaccine Dose for Year 1 & Year 2 Study Period
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day follow-up period after each vaccine dose for Year 1 & Year 2 study period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group
Number analyzed (Participants) | 876
Participants | 334

3. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs) During the 31-day Follow-up Period After Each Vaccine Dose for Year 3 & Year 4 Study Period
Description: as for outcome 2
Time Frame: During the 31-day follow-up period after each vaccine dose for Year 3 & Year 4 study period
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one dose of Rotarix vaccine administration documented and for whom data were available at Year 3 and Year 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group
Number analyzed (Participants) | 1052
Participants | 413

4. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs) During the 31-day Follow-up Period After Each Vaccine Dose for Year 5 Study Period
Description: as for outcome 2
Time Frame: During the 31 day follow-up period after each vaccine dose for Year 5 study period
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one dose of Rotarix vaccine administration documented and for whom data were available at Year 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group
Number analyzed (Participants) | 708
Participants | 254

5. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs) During the 31-day Follow-up Period After Each Vaccine Dose for Year 1 to Year 6 Study Period
Description: as for outcome 2
Time Frame: During the 31-day follow-up period after each vaccine dose for Year 1 to Year 6 study period
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one dose of Rotarix vaccine administration documented and for whom data were available for the Year 1 to Year 6 study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group
Number analyzed (Participants) | 3111
Participants | 1201

6. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) During the Post-marketing Study Period for Year 1 & Year 2 Study Period
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or were a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the post-marketing study period for Year 1 & Year 2 study period
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one dose of Rotarix vaccine administration documented for whom data were available at Year 1 and Year 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group
Number analyzed (Participants) | 876
Participants | 6

7. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) During the Post-marketing Study Period for Year 3 & Year 4 Study Period
Description: as for outcome 6
Time Frame: During the post-marketing study period for Year 3 & Year 4 study period
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one dose of Rotarix vaccine administration documented for whom data were available at Year 3 and Year 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group
Number analyzed (Participants) | 1052
Participants | 13

8. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) During the Post-marketing Study Period for Year 5 Study Period
Description: as for outcome 6
Time Frame: During the post-marketing study period for Year 5 study period
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one dose of Rotarix vaccine administration documented for whom data were available at Year 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group
Number analyzed (Participants) | 708
Participants | 4

9. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) During the Post-marketing Study Period for Year 1 to Year 6 Study Period
Description: as for outcome 6
Time Frame: During the post-marketing study period for Year 1 to Year 6 study period
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one dose of Rotarix vaccine administration documented and for whom data were available for Year 1 to Year 6 study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group
Number analyzed (Participants) | 3111
Participants | 26

ADVERSE EVENTS:
Time Frame: Serious adverse events: during Years 1, 2, 3, 4, 5 and 6 post-marketing study period. Systematically and non-systematically assessed frequent adverse events: during the 8-day and 31-day follow-up period after each vaccine dose, respectively.
Description: Classification for AEs was performed differently across the study period, according to MedDRA preferred terms until Year 4, and to World Health Organisation's Adverse Reactions Terminology (WHO ART) Dictionary for Year 5 and for the consolidated results from Year 1 to Year 6. The data presented within the Adverse Events section represent the consolidated results for Year 1 to Year 6 period.
Arm/Group | Rotarix Group
All-Cause Mortality (participants affected / at risk) | 0/3111
Serious Adverse Events (participants affected / at risk) | 26/3111
Other Adverse Events (participants affected / at risk) | 684/3111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=3111)
Ileus paralytic (Gastrointestinal disorders) | 1 — "Gastro-intestinal system disorders" SOC as per WHO-ART dictionary.
Colitis (Gastrointestinal disorders) | 1 — "Gastro-intestinal system disorders" SOC as per WHO-ART dictionary.
Otitis Media (Ear and labyrinth disorders) | 4 — "Resistance mechanism disorders" SOC as per WHO-ART dictionary.
Sepsis (Infections and infestations) | 1 — "Resistance mechanism disorders" SOC as per WHO-ART dictionary.
Gastroenteritis (Gastrointestinal disorders) | 3 — "Gastro-intestinal system disorders" SOC as per WHO-ART dictionary.
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 — "Respiratory system disorders" SOC as per WHO-ART dictionary.
Hydronephrosis (Renal and urinary disorders) | 1 — "Urinary System Disorders" SOC as per WHO-ART dictionary.
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1 — "Respiratory system disorders" SOC as per WHO-ART dictionary.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 — "Respiratory system disorders" SOC as per WHO-ART dictionary.
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 9 — "Respiratory system disorders" SOC as per WHO-ART dictionary.
Croup (Respiratory, thoracic and mediastinal disorders) | 1 — "Respiratory system disorders" SOC as per WHO-ART dictionary.
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 — "Respiratory system disorders" SOC as per WHO-ART dictionary.
Gastroenteritis viral (Gastrointestinal disorders) | 1 — "Gastro-intestinal system disorders" SOC as per WHO-ART dictionary.
Pneumonia viral (Respiratory, thoracic and mediastinal disorders) | 1 — "Respiratory system disorders" SOC as per WHO-ART dictionary.
Urinary tract infection (Renal and urinary disorders) | 3 — "Urinary System Disorders" SOC as per WHO-ART dictionary.
Fever (General disorders) | 1 — "Body as a whole - general disorders" SOC as per WHO-ART dictionary.
Cytomegalovirus Gastrointestinal Infection (Gastrointestinal disorders) | 1 — "Secondary items - events" SOC as per WHO-ART dictionary.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=3111)
Cough (Respiratory, thoracic and mediastinal disorders) | 204
Decreased appetite (Metabolism and nutrition disorders) | 259
Irritability (General disorders) | 405
Vomiting (Gastrointestinal disorders) | 200
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 268

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.